CLINICAL TRIAL: NCT04216550
Title: MR and Histopathology Images Based Prediction of Therapeutic Response of Apatinib in Recurrent Gliomas Using Artificial Intelligence
Brief Title: Prediction of Therapeutic Response of Apatinib in Recurrent Gliomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Zhenyu Zhang, Principal Investigator, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: GliomaAI-5
Record Dates: First submitted 2019-12-31; First posted 2020-01-02 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Recurrent Glioma
Keywords: Therapeutic responses; Radiological; Histopathology Imaging; Artificial intelligence; Apatinib
MeSH Terms: conditions — Glioma | interventions — apatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples With DNA — All participants have signed the informed consent. Fresh frozen tissues of participants are collected immediately after tumor resection and preserved in liquid nitrogen. Whole exome sequencing, RNA sequencing and proteomics are planed to be conducted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Apatinib: Apatinib 0.5g orally daily until the untolerable toxicities, disease progression or death
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 0.5g orally daily until the untolerable toxicities, disease progression or death

SUMMARY:
Apatinib, also known as YN968D1, is a small-molecule tyrosine kinase inhibitor (TKI) that selectively binds to and inhibits vascular endothelial growth factor receptor 2 (VEGFR-2). This study aims to collect clinical, radiological and histopathology imaging including detailed radiological data, survival data, clinical parameters, molecular pathology and images of HE slices in patients with recurrent gliomas whose are treated with Apatinib, for evaluating the efficacy and safety of Apatinib. Moreover, by leveraging artificial intelligence, this study seeks to construct and refine MR and histopathology imaging based algorithms that are able to predict the responses to Apatinib of patients with recurrent gliomas.

DETAILED DESCRIPTION:
Effective treatment for recurrent gliomas is still challenging. Malignant gliomas are considered to be one of the most angiogenic cancers and are mostly sustained by vascular endothelial growth factor (VEGF) signaling via its endothelial tyrosine kinase receptor VEGF receptor 2 (VEGFR-2). Apatinib, also known as YN968D1, is a small-molecule tyrosine kinase inhibitor (TKI) that selectively binds to and inhibits VEGFR-2. Apatinib has been demonstrated as monotherapy that prolongs OS in patients with gastric cancers after two or more lines of chemotherapy with moderate, reversible, and easily managed adverse effects. This study aims to collect clinical, radiological and histopathology imaging including detailed radiological data, survival data, clinical parameters, molecular pathology and images of HE slices in patients with recurrent gliomas whose are treated with Apatinib, for evaluating the efficacy and safety of Apatinib. Moreover, by leveraging artificial intelligence, this study also seeks to construct and refine MR and histopathology imaging based algorithms that are able to predict the responses to Apatinib of patients with recurrent gliomas. The creation of a registry for patients with recurrent gliomas treated by Apatinib with detailed survival data, radiological data, histopathology image data and with sufficient sample size for artificial intelligence provides opportunities for personalized prediction of responses to Apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with histologically-confirmed WHO Grade II-IV gliomas which have recurrent or progressive conditions.
2. With measurable or evaluable disease defined by RANO criteria by MRI scan.
3. Eastern Cooperative Oncology Group Performance Status (ECOG P.S.) of ≤ 2
4. Life expectancy ≥3 months.
5. No evidence of serious cardiopulmonary function damage, postoperative complication and hemorrhage on the baseline.
6. No history of serious hypertension disease.
7. Patients have adequate organ function as defined by the following criteria:

   * Hemoglobin (HGB) ≥90g/L
   * Absolute neutrophil count (ANC) ≥1.5×109/L
   * White blood cell (WBC) ≥3.0×109/L
   * Platelet count ≥80×109/L
   * Alanine aminotransferase(ALT) and Aspartate aminotransferase (AST) of ≤2.5 upper normal limitation (UNL) or ≤5 UNL in case of liver metastasis
   * Creatinine (Cr) of ≤1.25 UNL or creatinine clearance(Ccr) > 45 ml/min.
8. With written informed consent signed voluntarily by patients themselves.

Exclusion Criteria:

1. Patients with age<18 or >90 years.
2. Pregnant or lactating women.
3. Inadequately controlled hypertension (defined as systolic blood pressure > 140 and/or diastolic blood pressure > 90 mmHg on antihypertensive medications).
4. New York Heart Association (NYHA) Grade II or greater congestive heart failure.
5. Factors that could have an effect on oral medication.
6. Abnormal Coagulation (international normalized ratio>1.5, prothrombin time>UNL+4s,activated partial thromboplastin time>1.5 UNL), with tendency of bleeding.
7. Currently receive thrombolytic and anticoagulation therapy
8. History of pneumorrhagia(CTCAE grade ≥2 ) or other parts hemorrhage(CTCAE grade ≥3 ) within 4 weeks prior to treatment.
9. History of artery thrombosis and phlebothrombosis, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism, within 6 month prior to treatment.
10. Medical history of clinically significant thrombosis (bleeding or clotting disorder), excluding warfarin(1mg po qd) and aspirin(80-100mg po qd) for prevention under INR≤1.5.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are all received anti-angiogenesis drug (Apatinib) in the First Affiliated Hospital of Zhengzhou University.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes of Response to Treatment | From enrollment to progression of disease. Estimated about 6 months
  Response were evaluated with Response Assessment in Neuro-Oncology (RANO) criteria every 1 month after treament.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From enrollment to progression of disease. Estimated about 6 months.
  The length of time from enrollment until the time of progression of disease (PFS, progression-free survival)
Overall Survival (OS) | From enrollment to death of patients. Estimated about 1 year.
  The length of time from enrollment until the time of death (OS, overall survival)
Incidence of treatment-related adverse events | Time Frame: 0 to 1 year
  The incidence of treatment-related adverse events were graded with the use of the National Cancer Institute Common Terminology Criteria for Adverse Events, version 4.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided